CLINICAL TRIAL: NCT03333759
Title: Treatment of Atrophic Facial Acne Scars With Er:YAG Laser Examined Under Optical Coherence Tomography
Brief Title: Treatment of Acne Scars With Erbium:Yttrium Aluminum Garnet (Er:YAG) Laser Examined Under OCT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult recruiting participants
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Keyvan Nouri, Doctor of Medicine, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20170490
Record Dates: First submitted 2017-08-01; First posted 2017-11-07 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Acne Vulgaris
Keywords: laser; Er:YAG laser; acne; acne vulgaris; optical coherence tomography
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Laser Treatment (Experimental): Patients will receive one laser treatment (week 0) with the Erbium YAG laser at a 2940nm wavelength (Alma - Harmony XL Laser) and parameters corresponding with their acne scar severity. They will then return to the clinic 1, 4 and 8 weeks (7, 30, and 56 days + 7 days) after the treatment for their scars to be evaluated under optical coherence tomography.
  Laser parameters are as follows:
  iPixelEr 2940nm Erbium:YAG Module: mild scars: 7 by 7 (7X7) mm tip, energy 1400-1600 millijoules/P (mJ), pulse energy 5 Hz, 2-6 stacks, pulse mode L, 2-3 passes, 10% overlap moderate scars: 7X7 mm tip, energy 1600-1800 mJ/P, pulse energy 5 Hz, 2-6 stacks, pulse mode L, 2-3 passes, 10% overlap severe scars: 7X7 mm tip, 1800-2000 mJ/P, pulse energy 5 Hz, 2-6 stacks, pulse mode L, 2-3 passes, 10% overlap
  Interventions: Device: Alma - Harmony XL Laser

INTERVENTIONS:
Device: Alma - Harmony XL Laser — The Erbium YAG laser at a 2940nm wavelength is used for ablative laser resurfacing as well as treating acne scars.
  Other Names: Modified Alma Laser Harmony Neodymium-Doped Yttrium Aluminium Garnet (Nd:YAG) Module

SUMMARY:
This study is examining the effects of the 2940 nm Er:YAG on atrophic facial acne scars under optical coherence tomography in terms of blood flow, vessel shape, skin roughness, collagen content, and epidermal thickness.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should be 18-90 years of age
2. Patients should have Fitzpatrick skin types of I-III
3. Patients should have at least mild acne

Exclusion Criteria:

1. The patient should not be receiving any additional systemic, topical, or intralesional treatment of the scars during the study
2. Pregnant or lactating females
3. Fitzpatrick skin type of IV-VI
4. A history of keloids or hypertrophic scars
5. Scleroderma
6. Photosensitivity
7. Botulinum toxin injection, facial laser resurfacing, chemical peels, fillers, or usage of oral retinoid within the last 6 months
8. Subjects with a known history of herpes simplex

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in blood flow | During 8 weeks
  Optical coherence tomography (OCT) will be used to quantitatively measure changes in facial atrophic acne scars in terms of blood flow (proportion of signals with strong dynamic signal (%)/depth (mm)).
Change in epidermal thickness | During 8 weeks
  Optical coherence tomography (OCT) will be used to quantitatively measure changes in facial atrophic acne scars in terms of epidermal thickness (mm).
Change in collagen content | During 8 weeks
  OCT will be used to qualitatively measure changes in facial atrophic acne scars in terms of collagen content. Collagen content will be measured in terms of brightness of OCT scan. Areas of skin that contain collagen tend to be brighter (more white in color) whereas areas with less collagen content tend to be darker.
Change in skin roughness | During 8 weeks
  OCT will be used to quantitatively measure changes in facial atrophic acne scars in terms of skin roughness (µm).

SECONDARY OUTCOMES:
The Patient Scar Assessment Scale | During 8 weeks
  Scale (1-10) used to qualitatively monitor treatment and changes in scars by the patient.
The Observer Scar Assessment Scale | During 8 weeks
  Scale (1-10) used to qualitatively monitor treatment and changes in scars by the dermatologist.

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Nouri, MD, Principal Investigator — University of Miami
Locations (1):
- Sylvester Comprehensive Cancer Center, Miami, Florida, United States